CLINICAL TRIAL: NCT00005260
Title: Mechanisms Underlying Psychosocial Associations With Ischemic Heart Disease (Kuopio)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1143; R01HL044199 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2005-07

CONDITIONS: Cardiovascular Diseases; Carotid Artery Diseases; Arrhythmia; Myocardial Ischemia; Thrombosis; Heart Diseases; Atherosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Carotid Artery Diseases; Arrhythmias, Cardiac; Myocardial Ischemia; Thrombosis; Heart Diseases; Atherosclerosis

SUMMARY:
To examine the relationships among psychosocial factors and carotid atherosclerosis, myocardial ischemia, arrhythmias, and thrombosis.

DETAILED DESCRIPTION:
BACKGROUND:

Considerable interest and controversy exist concerning the role of psychosocial factors in the pathogenesis of ischemic heart disease. Studies of the prevalence, incidence, and mortality from ischemic heart disease have implicated socioeconomic status, job strain, Type A behavior, hostility, social support, and other variables.

The study used baseline data previously collected as part of the Kuopio Ischemic Heart Disease Risk Factor Study conducted in eastern Finland by the Research Institute of Public Health and the Research Institute of Exercise Medicine, both in Kuopio, and the Finnish National Public Health Institute in Helsinki. The area of eastern Finland lies within the area of greatest morbidity and mortality from ischemic heart disease in Finland, was part of the reference area for the evaluation of the North Karelia Project, and is part of the World Health Organization MONICA project.

DESIGN NARRATIVE:

The study was longitudinal in design. Physical examinations were conducted at baseline and information collected on behavioral risk factors, medical history, and medications. Evaluations included a maximal exercise tolerance test, four day supervised food recordings, a broad set of hematological and chemical tests from fasting venous blood and two 24-hour urine samples. Holter monitoring and ultrasonography of the carotid arteries were performed in Cohort II only. Psychosocial measures included social support and network participation, socioeconomic status, job strain, Type A behavior pattern, and John Henryism. All members of Cohort II were re-examined three years post-baseline. Cohort I members were not re-examined because they did not undergo Holter monitoring and ultrasonography. Prevalence and ischemic heart disease incidence analyses were performed using both cohorts. Baseline psychosocial factors were examined in relation to study endpoints which included extent of carotid atherosclerosis, presence of ischemia on exercise, presence of arrhythmias, tendency toward blood clotting, four year progression of atherosclerosis, and incidence of fatal and non-fatal ischemic heart disease.

The study was renewed in 1997. Data from a baseline examination, a four-year re-examination, and a proposed one-year re-examination of ultrasonographically assessed carotid and femoral atherosclerosis, and surveillance for myocardial infarctions and other outcomes, will be used to examine the progression or incidence of these outcomes in relation to changes in behavioral, psychosocial and socioeconomic factors. It will also be possible to see to to what extent the input of these behavioral, psychosocial and socioeconomic factors on cardiovascular disease (CVD) in 1,600 men and women is mediated by lipid peroxidation, hemostatic factors, and cardiovascular reactivity. Finally, the investigators state that this will be the first population-based epidemiologic study to examine the association between a carefully developed set of measures of cardiovascular reactivity to stress and the progression of carotid atherosclerosis, risk of myocardial infarction and death, and development of hypertension. The cohorts had previously been all male. Women were added when the study was renewed in FY 1997.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1990-07; Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Kaplan — University of Michigan

REFERENCES:
- [Background] Wilson TW, Cohen RD, Lachenbruch PA, Wu M, Kaplan GA, Salonen JT. Is the relationship between supine blood pressure and postural changes in blood pressure artefactual? Results from the Kuopio Ischemic Heart Disease Risk Factor Study. J Hypertens. 1995 Apr;13(4):421-6. PMID 7629402
- [Background] Lynch JW, Everson SA, Kaplan GA, Salonen R, Salonen JT. Does low socioeconomic status potentiate the effects of heightened cardiovascular responses to stress on the progression of carotid atherosclerosis? Am J Public Health. 1998 Mar;88(3):389-94. doi: 10.2105/ajph.88.3.389. PMID 9518969
- [Background] Salonen JT, Lakka TA, Lakka HM, Valkonen VP, Everson SA, Kaplan GA. Hyperinsulinemia is associated with the incidence of hypertension and dyslipidemia in middle-aged men. Diabetes. 1998 Feb;47(2):270-5. doi: 10.2337/diab.47.2.270. PMID 9519724
- [Background] Kamarck TW, Everson SA, Kaplan GA, Manuck SB, Jennings JR, Salonen R, Salonen JT. Exaggerated blood pressure responses during mental stress are associated with enhanced carotid atherosclerosis in middle-aged Finnish men: findings from the Kuopio Ischemic Heart Disease Study. Circulation. 1997 Dec 2;96(11):3842-8. doi: 10.1161/01.cir.96.11.3842. PMID 9403606
- [Background] Kauhanen J, Kaplan GA, Goldberg DE, Salonen JT. Beer binging and mortality: results from the Kuopio ischaemic heart disease risk factor study, a prospective population based study. BMJ. 1997 Oct 4;315(7112):846-51. doi: 10.1136/bmj.315.7112.846. PMID 9353504
- [Background] Lynch J, Helmrich SP, Lakka TA, Kaplan GA, Cohen RD, Salonen R, Salonen JT. Moderately intense physical activities and high levels of cardiorespiratory fitness reduce the risk of non-insulin-dependent diabetes mellitus in middle-aged men. Arch Intern Med. 1996 Jun 24;156(12):1307-14. PMID 8651839
- [Background] Everson SA, Kaplan GA, Goldberg DE, Salonen R, Salonen JT. Hopelessness and 4-year progression of carotid atherosclerosis. The Kuopio Ischemic Heart Disease Risk Factor Study. Arterioscler Thromb Vasc Biol. 1997 Aug;17(8):1490-5. doi: 10.1161/01.atv.17.8.1490. PMID 9301625
- [Background] Everson SA, Kauhanen J, Kaplan GA, Goldberg DE, Julkunen J, Tuomilehto J, Salonen JT. Hostility and increased risk of mortality and acute myocardial infarction: the mediating role of behavioral risk factors. Am J Epidemiol. 1997 Jul 15;146(2):142-52. doi: 10.1093/oxfordjournals.aje.a009245. PMID 9230776
- [Background] Lynch J, Krause N, Kaplan GA, Salonen R, Salonen JT. Workplace demands, economic reward, and progression of carotid atherosclerosis. Circulation. 1997 Jul 1;96(1):302-7. doi: 10.1161/01.cir.96.1.302. PMID 9236449
- [Background] Jennings JR, Kamarck T, Manuck S, Everson SA, Kaplan G, Salonen JT. Aging or disease? Cardiovascular reactivity in Finnish men over the middle years. Psychol Aging. 1997 Jun;12(2):225-38. doi: 10.1037//0882-7974.12.2.225. PMID 9189982
- [Background] Lynch J, Krause N, Kaplan GA, Tuomilehto J, Salonen JT. Workplace conditions, socioeconomic status, and the risk of mortality and acute myocardial infarction: the Kuopio Ischemic Heart Disease Risk Factor Study. Am J Public Health. 1997 Apr;87(4):617-22. doi: 10.2105/ajph.87.4.617. PMID 9146441
- [Background] Kauhanen J, Kaplan GA, Goldberg DD, Cohen RD, Lakka TA, Salonen JT. Frequent hangovers and cardiovascular mortality in middle-aged men. Epidemiology. 1997 May;8(3):310-4. doi: 10.1097/00001648-199705000-00014. PMID 9115028
- [Background] Tuomainen TP, Nyyssonen K, Salonen R, Tervahauta A, Korpela H, Lakka T, Kaplan GA, Salonen JT. Body iron stores are associated with serum insulin and blood glucose concentrations. Population study in 1,013 eastern Finnish men. Diabetes Care. 1997 Mar;20(3):426-8. doi: 10.2337/diacare.20.3.426. PMID 9051399
- [Background] Lynch JW, Kaplan GA, Salonen JT. Why do poor people behave poorly? Variation in adult health behaviours and psychosocial characteristics by stages of the socioeconomic lifecourse. Soc Sci Med. 1997 Mar;44(6):809-19. doi: 10.1016/s0277-9536(96)00191-8. PMID 9080564
- [Background] Kauhanen J, Kaplan GA, Cohen RD, Julkunen J, Salonen JT. Alexithymia and risk of death in middle-aged men. J Psychosom Res. 1996 Dec;41(6):541-9. doi: 10.1016/s0022-3999(96)00226-7. PMID 9032717
- [Background] Lynch J, Kaplan GA, Salonen R, Salonen JT. Socioeconomic status and progression of carotid atherosclerosis. Prospective evidence from the Kuopio Ischemic Heart Disease Risk Factor Study. Arterioscler Thromb Vasc Biol. 1997 Mar;17(3):513-9. doi: 10.1161/01.atv.17.3.513. PMID 9102170
- [Background] Everson SA, Lynch JW, Chesney MA, Kaplan GA, Goldberg DE, Shade SB, Cohen RD, Salonen R, Salonen JT. Interaction of workplace demands and cardiovascular reactivity in progression of carotid atherosclerosis: population based study. BMJ. 1997 Feb 22;314(7080):553-8. doi: 10.1136/bmj.314.7080.553. PMID 9055713
- [Background] Rasanen J, Kauhanen J, Lakka TA, Kaplan GA, Salonen JT. Religious affiliation and all-cause mortality: a prospective population study in middle-aged men in eastern Finland. Int J Epidemiol. 1996 Dec;25(6):1244-9. doi: 10.1093/ije/25.6.1244. PMID 9027531
- [Background] Lynch JW, Kaplan GA, Cohen RD, Tuomilehto J, Salonen JT. Do cardiovascular risk factors explain the relation between socioeconomic status, risk of all-cause mortality, cardiovascular mortality, and acute myocardial infarction? Am J Epidemiol. 1996 Nov 15;144(10):934-42. doi: 10.1093/oxfordjournals.aje.a008863. PMID 8916504
- [Background] Everson SA, Kaplan GA, Goldberg DE, Salonen JT. Anticipatory blood pressure response to exercise predicts future high blood pressure in middle-aged men. Hypertension. 1996 May;27(5):1059-64. doi: 10.1161/01.hyp.27.5.1059. PMID 8621197
- [Background] Salonen JT, Nyyssonen K, Tuomainen TP, Maenpaa PH, Korpela H, Kaplan GA, Lynch J, Helmrich SP, Salonen R. Increased risk of non-insulin dependent diabetes mellitus at low plasma vitamin E concentrations: a four year follow up study in men. BMJ. 1995 Oct 28;311(7013):1124-7. doi: 10.1136/bmj.311.7013.1124. PMID 7580706
- [Background] Lynch J, Kaplan GA, Salonen R, Cohen RD, Salonen JT. Socioeconomic status and carotid atherosclerosis. Circulation. 1995 Oct 1;92(7):1786-92. doi: 10.1161/01.cir.92.7.1786. PMID 7671362
- [Background] Kaplan GA, Wilson TW, Cohen RD, Kauhanen J, Wu M, Salonen JT. Social functioning and overall mortality: prospective evidence from the Kuopio Ischemic Heart Disease Risk Factor Study. Epidemiology. 1994 Sep;5(5):495-500. PMID 7986863
- [Background] Lynch JW, Kaplan GA, Cohen RD, Kauhanen J, Wilson TW, Smith NL, Salonen JT. Childhood and adult socioeconomic status as predictors of mortality in Finland. Lancet. 1994 Feb 26;343(8896):524-7. doi: 10.1016/s0140-6736(94)91468-0. PMID 7906766
- [Background] Kauhanen J, Kaplan GA, Cohen RD, Salonen R, Salonen JT. Alexithymia may influence the diagnosis of coronary heart disease. Psychosom Med. 1994 May-Jun;56(3):237-44. doi: 10.1097/00006842-199405000-00010. PMID 8084970
- [Background] Wilson TW, Kaplan GA, Kauhanen J, Cohen RD, Wu M, Salonen R, Salonen JT. Association between plasma fibrinogen concentration and five socioeconomic indices in the Kuopio Ischemic Heart Disease Risk Factor Study. Am J Epidemiol. 1993 Feb 1;137(3):292-300. doi: 10.1093/oxfordjournals.aje.a116676. PMID 8452137
- [Background] Kauhanen J, Hallikainen T, Tuomainen TP, Koulu M, Karvonen MK, Salonen JT, Tiihonen J. Association between the functional polymorphism of catechol-O-methyltransferase gene and alcohol consumption among social drinkers. Alcohol Clin Exp Res. 2000 Feb;24(2):135-9. PMID 10698363
- [Background] Everson SA, Kaplan GA, Goldberg DE, Salonen JT. Hypertension incidence is predicted by high levels of hopelessness in Finnish men. Hypertension. 2000 Feb;35(2):561-7. doi: 10.1161/01.hyp.35.2.561. PMID 10679498
- [Background] Salonen JT, Seppanen K, Lakka TA, Salonen R, Kaplan GA. Mercury accumulation and accelerated progression of carotid atherosclerosis: a population-based prospective 4-year follow-up study in men in eastern Finland. Atherosclerosis. 2000 Feb;148(2):265-73. doi: 10.1016/s0021-9150(99)00272-5. PMID 10657561
- [Background] Kaplan GA, Lynch JW. Socioeconomic considerations in the primordial prevention of cardiovascular disease. Prev Med. 1999 Dec;29(6 Pt 2):S30-5. doi: 10.1006/pmed.1999.0540. PMID 10641815
- [Background] Vanharanta M, Voutilainen S, Lakka TA, van der Lee M, Adlercreutz H, Salonen JT. Risk of acute coronary events according to serum concentrations of enterolactone: a prospective population-based case-control study. Lancet. 1999 Dec 18-25;354(9196):2112-5. doi: 10.1016/S0140-6736(99)05031-X. PMID 10609816
- [Background] Kauhanen J, Kaplan GA, Goldberg DE, Salonen R, Salonen JT. Pattern of alcohol drinking and progression of atherosclerosis. Arterioscler Thromb Vasc Biol. 1999 Dec;19(12):3001-6. doi: 10.1161/01.atv.19.12.3001. PMID 10591681
- [Background] Tuomainen TP, Kontula K, Nyyssonen K, Lakka TA, Helio T, Salonen JT. Increased risk of acute myocardial infarction in carriers of the hemochromatosis gene Cys282Tyr mutation : a prospective cohort study in men in eastern Finland. Circulation. 1999 Sep 21;100(12):1274-9. doi: 10.1161/01.cir.100.12.1274. PMID 10491370
- [Background] Salonen JT, Malin R, Tuomainen TP, Nyyssonen K, Lakka TA, Lehtimaki T. Polymorphism in high density lipoprotein paraoxonase gene and risk of acute myocardial infarction in men: prospective nested case-control study. BMJ. 1999 Aug 21;319(7208):487-9; discussion 490. doi: 10.1136/bmj.319.7208.487. No abstract available. PMID 10454401
- [Background] Lakka TA, Salonen R, Kaplan GA, Salonen JT. Blood pressure and the progression of carotid atherosclerosis in middle-aged men. Hypertension. 1999 Jul;34(1):51-6. doi: 10.1161/01.hyp.34.1.51. PMID 10406823
- [Background] Everson SA, Kaplan GA, Goldberg DE, Lakka TA, Sivenius J, Salonen JT. Anger expression and incident stroke: prospective evidence from the Kuopio ischemic heart disease study. Stroke. 1999 Mar;30(3):523-8. doi: 10.1161/01.str.30.3.523. PMID 10066846
- [Background] Everson SA, Goldberg DE, Kaplan GA, Julkunen J, Salonen JT. Anger expression and incident hypertension. Psychosom Med. 1998 Nov-Dec;60(6):730-5. doi: 10.1097/00006842-199811000-00014. PMID 9847033
- [Background] Everson SA, Goldberg DE, Helmrich SP, Lakka TA, Lynch JW, Kaplan GA, Salonen JT. Weight gain and the risk of developing insulin resistance syndrome. Diabetes Care. 1998 Oct;21(10):1637-43. doi: 10.2337/diacare.21.10.1637. PMID 9773723
- [Background] Salonen JT, Tuomainen TP, Nyyssonen K, Lakka HM, Punnonen K. Relation between iron stores and non-insulin dependent diabetes in men: case-control study. BMJ. 1998 Sep 12;317(7160):727. doi: 10.1136/bmj.317.7160.727. No abstract available. PMID 9732340
- [Background] Salonen JT. Excessive intake of iron and mercury in cardiovascular disease. Bibl Nutr Dieta. 1998;(54):112-26. doi: 10.1159/000059452. No abstract available. PMID 9597177
- [Background] Lakka TA, Laukkanen JA, Rauramaa R, Salonen R, Lakka HM, Kaplan GA, Salonen JT. Cardiorespiratory fitness and the progression of carotid atherosclerosis in middle-aged men. Ann Intern Med. 2001 Jan 2;134(1):12-20. doi: 10.7326/0003-4819-134-1-200101020-00008. PMID 11187415
- [Background] Lakka TA, Lakka HM, Salonen R, Kaplan GA, Salonen JT. Abdominal obesity is associated with accelerated progression of carotid atherosclerosis in men. Atherosclerosis. 2001 Feb 1;154(2):497-504. doi: 10.1016/s0021-9150(00)00514-1. PMID 11166785
- [Background] Lakka HM, Oksanen L, Tuomainen TP, Kontula K, Salonen JT. The common pentanucleotide polymorphism of the 3'-untranslated region of the leptin receptor gene is associated with serum insulin levels and the risk of type 2 diabetes in non-diabetic men: a prospective case-control study. J Intern Med. 2000 Jul;248(1):77-83. doi: 10.1046/j.1365-2796.2000.00696.x. PMID 10947884
- [Background] Krause N, Lynch JW, Kaplan GA, Cohen RD, Salonen R, Salonen JT. Standing at work and progression of carotid atherosclerosis. Scand J Work Environ Health. 2000 Jun;26(3):227-36. doi: 10.5271/sjweh.536. PMID 10901115
- [Background] Kauhanen J, Karvonen MK, Pesonen U, Koulu M, Tuomainen TP, Uusitupa MI, Salonen JT. Neuropeptide Y polymorphism and alcohol consumption in middle-aged men. Am J Med Genet. 2000 Jul 17;93(2):117-21. doi: 10.1002/1096-8628(20000717)93:23.0.co;2-#. PMID 10869113
- [Background] Salonen JT, Tuomainen TP, Kontula K. Role of C282Y mutation in haemochromatosis gene in development of type 2 diabetes in healthy men: prospective cohort study. BMJ. 2000 Jun 24;320(7251):1706-7. doi: 10.1136/bmj.320.7251.1706. No abstract available. PMID 10864547
- [Background] Helkala EL, Lakka T, Vanhanen M, Tuomainen TP, Ehnholm C, Kaplan GA, Salonen JT. Associations between apolipoprotein E phenotype, glucose metabolism and cognitive function in men. An explorative study in a population sample. Diabet Med. 2001 Dec;18(12):991-7. doi: 10.1046/j.0742-3071.2001.00588.x. PMID 11903399
- [Background] Turrell G, Lynch JW, Kaplan GA, Everson SA, Helkala EL, Kauhanen J, Salonen JT. Socioeconomic position across the lifecourse and cognitive function in late middle age. J Gerontol B Psychol Sci Soc Sci. 2002 Jan;57(1):S43-51. doi: 10.1093/geronb/57.1.s43. PMID 11773232
- [Background] Everson SA, Lynch JW, Kaplan GA, Lakka TA, Sivenius J, Salonen JT. Stress-induced blood pressure reactivity and incident stroke in middle-aged men. Stroke. 2001 Jun;32(6):1263-70. doi: 10.1161/01.str.32.6.1263. PMID 11387485
- [Background] Kaplan GA, Turrell G, Lynch JW, Everson SA, Helkala EL, Salonen JT. Childhood socioeconomic position and cognitive function in adulthood. Int J Epidemiol. 2001 Apr;30(2):256-63. doi: 10.1093/ije/30.2.256. PMID 11369724
- [Background] Vanharanta M, Voutilainen S, Rissanen TH, Adlercreutz H, Salonen JT. Risk of cardiovascular disease-related and all-cause death according to serum concentrations of enterolactone: Kuopio Ischaemic Heart Disease Risk Factor Study. Arch Intern Med. 2003 May 12;163(9):1099-104. doi: 10.1001/archinte.163.9.1099. PMID 12742810
- [Background] Lakka HM, Laaksonen DE, Lakka TA, Niskanen LK, Kumpusalo E, Tuomilehto J, Salonen JT. The metabolic syndrome and total and cardiovascular disease mortality in middle-aged men. JAMA. 2002 Dec 4;288(21):2709-16. doi: 10.1001/jama.288.21.2709. PMID 12460094
- [Background] Laaksonen DE, Lakka HM, Niskanen LK, Kaplan GA, Salonen JT, Lakka TA. Metabolic syndrome and development of diabetes mellitus: application and validation of recently suggested definitions of the metabolic syndrome in a prospective cohort study. Am J Epidemiol. 2002 Dec 1;156(11):1070-7. doi: 10.1093/aje/kwf145. PMID 12446265
- [Background] Lakka HM, Salonen JT, Tuomilehto J, Kaplan GA, Lakka TA. Obesity and weight gain are associated with increased incidence of hyperinsulinemia in non-diabetic men. Horm Metab Res. 2002 Sep;34(9):492-8. doi: 10.1055/s-2002-34788. PMID 12384825
- [Background] Everson SA, Maty SC, Lynch JW, Kaplan GA. Epidemiologic evidence for the relation between socioeconomic status and depression, obesity, and diabetes. J Psychosom Res. 2002 Oct;53(4):891-5. doi: 10.1016/s0022-3999(02)00303-3. PMID 12377299
- [Background] Laaksonen DE, Lakka TA, Lakka HM, Nyyssonen K, Rissanen T, Niskanen LK, Salonen JT. Serum fatty acid composition predicts development of impaired fasting glycaemia and diabetes in middle-aged men. Diabet Med. 2002 Jun;19(6):456-64. doi: 10.1046/j.1464-5491.2002.00707.x. PMID 12060056
- [Background] Kurl S, Tuomainen TP, Laukkanen JA, Nyyssonen K, Lakka T, Sivenius J, Salonen JT. Plasma vitamin C modifies the association between hypertension and risk of stroke. Stroke. 2002 Jun;33(6):1568-73. doi: 10.1161/01.str.0000017220.78722.d7. PMID 12052992
- [Background] Harper S, Lynch J, Hsu WL, Everson SA, Hillemeier MM, Raghunathan TE, Salonen JT, Kaplan GA. Life course socioeconomic conditions and adult psychosocial functioning. Int J Epidemiol. 2002 Apr;31(2):395-403. PMID 11980802
- [Background] Lakka HM, Lakka TA, Tuomilehto J, Salonen JT. Abdominal obesity is associated with increased risk of acute coronary events in men. Eur Heart J. 2002 May;23(9):706-13. doi: 10.1053/euhj.2001.2889. PMID 11977996
- [Background] Laaksonen DE, Nyyssonen K, Niskanen L, Rissanen TH, Salonen JT. Prediction of cardiovascular mortality in middle-aged men by dietary and serum linoleic and polyunsaturated fatty acids. Arch Intern Med. 2005 Jan 24;165(2):193-9. doi: 10.1001/archinte.165.2.193. PMID 15668366
- [Background] Tolmunen T, Hintikka J, Voutilainen S, Ruusunen A, Alfthan G, Nyyssonen K, Viinamaki H, Kaplan GA, Salonen JT. Association between depressive symptoms and serum concentrations of homocysteine in men: a population study. Am J Clin Nutr. 2004 Dec;80(6):1574-8. doi: 10.1093/ajcn/80.6.1574. PMID 15585771
- [Background] Laukkanen JA, Kurl S, Salonen R, Lakka TA, Rauramaa R, Salonen JT. Systolic blood pressure during recovery from exercise and the risk of acute myocardial infarction in middle-aged men. Hypertension. 2004 Dec;44(6):820-5. doi: 10.1161/01.HYP.0000148460.95060.f2. Epub 2004 Nov 8. PMID 15534077
- [Background] Niskanen L, Laaksonen DE, Nyyssonen K, Punnonen K, Valkonen VP, Fuentes R, Tuomainen TP, Salonen R, Salonen JT. Inflammation, abdominal obesity, and smoking as predictors of hypertension. Hypertension. 2004 Dec;44(6):859-65. doi: 10.1161/01.HYP.0000146691.51307.84. Epub 2004 Oct 18. PMID 15492131
- [Background] Tolmunen T, Hintikka J, Ruusunen A, Voutilainen S, Tanskanen A, Valkonen VP, Viinamaki H, Kaplan GA, Salonen JT. Dietary folate and the risk of depression in Finnish middle-aged men. A prospective follow-up study. Psychother Psychosom. 2004 Nov-Dec;73(6):334-9. doi: 10.1159/000080385. PMID 15479987
- [Background] Laukkanen JA, Laaksonen DE, Niskanen L, Pukkala E, Hakkarainen A, Salonen JT. Metabolic syndrome and the risk of prostate cancer in Finnish men: a population-based study. Cancer Epidemiol Biomarkers Prev. 2004 Oct;13(10):1646-50. PMID 15466982
- [Background] Jennings JR, Kamarck TW, Everson-Rose SA, Kaplan GA, Manuck SB, Salonen JT. Exaggerated blood pressure responses during mental stress are prospectively related to enhanced carotid atherosclerosis in middle-aged Finnish men. Circulation. 2004 Oct 12;110(15):2198-203. doi: 10.1161/01.CIR.0000143840.77061.E9. Epub 2004 Sep 27. PMID 15451789
- [Background] Laukkanen JA, Kurl S, Salonen R, Rauramaa R, Salonen JT. The predictive value of cardiorespiratory fitness for cardiovascular events in men with various risk profiles: a prospective population-based cohort study. Eur Heart J. 2004 Aug;25(16):1428-37. doi: 10.1016/j.ehj.2004.06.013. PMID 15321701
- [Background] Laaksonen DE, Niskanen L, Nyyssonen K, Punnonen K, Tuomainen TP, Valkonen VP, Salonen R, Salonen JT. C-reactive protein and the development of the metabolic syndrome and diabetes in middle-aged men. Diabetologia. 2004 Aug;47(8):1403-10. doi: 10.1007/s00125-004-1472-x. Epub 2004 Jul 28. PMID 15309290
- [Background] Laaksonen DE, Laukkanen JA, Niskanen L, Nyyssonen K, Rissanen TH, Voutilainen S, Pukkala E, Hakkarainen A, Salonen JT. Serum linoleic and total polyunsaturated fatty acids in relation to prostate and other cancers: a population-based cohort study. Int J Cancer. 2004 Sep 1;111(3):444-50. doi: 10.1002/ijc.11614. PMID 15221975
- [Background] Laaksonen DE, Niskanen L, Punnonen K, Nyyssonen K, Tuomainen TP, Valkonen VP, Salonen R, Salonen JT. Testosterone and sex hormone-binding globulin predict the metabolic syndrome and diabetes in middle-aged men. Diabetes Care. 2004 May;27(5):1036-41. doi: 10.2337/diacare.27.5.1036. PMID 15111517
- [Background] Fan YM, Salonen JT, Koivu TA, Tuomainen TP, Nyyssonen K, Lakka TA, Salonen R, Seppanen K, Nikkari ST, Tahvanainen E, Lehtimaki T. Hepatic lipase C-480T polymorphism modifies the effect of HDL cholesterol on the risk of acute myocardial infarction in men: a prospective population based study. J Med Genet. 2004 Mar;41(3):e28. doi: 10.1136/jmg.2003.010652. No abstract available. PMID 14985399
- [Background] Laaksonen DE, Niskanen L, Punnonen K, Nyyssonen K, Tuomainen TP, Salonen R, Rauramaa R, Salonen JT. Sex hormones, inflammation and the metabolic syndrome: a population-based study. Eur J Endocrinol. 2003 Dec;149(6):601-8. doi: 10.1530/eje.0.1490601. PMID 14641004
- [Background] Salonen JT. Liver damage and protective effect of high density lipoprotein cholesterol. BMJ. 2003 Nov 8;327(7423):1082-3. doi: 10.1136/bmj.327.7423.1082. PMID 14604929
- [Background] Kurl S, Laukkanen JA, Rauramaa R, Lakka TA, Sivenius J, Salonen JT. Cardiorespiratory fitness and the risk for stroke in men. Arch Intern Med. 2003 Jul 28;163(14):1682-8. doi: 10.1001/archinte.163.14.1682. PMID 12885683
- [Background] Kurl S, Laukkanen JA, Tuomainen TP, Rauramaa R, Lakka TA, Salonen R, Eranen J, Sivenius J, Salonen JT. Association of exercise-induced, silent ST-segment depression with the risk of stroke and cardiovascular diseases in men. Stroke. 2003 Jul;34(7):1760-5. doi: 10.1161/01.STR.0000078564.46376.0A. Epub 2003 Jun 26. PMID 12829872
- [Background] Krause N, Lynch J, Kaplan GA, Cohen RD, Goldberg DE, Salonen JT. Predictors of disability retirement. Scand J Work Environ Health. 1997 Dec;23(6):403-13. doi: 10.5271/sjweh.262. PMID 9476803